CLINICAL TRIAL: NCT01742728
Title: Oxidative Stress in Community-dwelling Adults
Brief Title: Nagasaki and Tokushima
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Tokushima (Other)
Responsible Party: Principal Investigator, Naofumi Tamaki, oxidative stress and periodontitis, University of Tokushima
Other Study IDs: goto2012
Record Dates: First submitted 2012-11-28; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Periodontitis
Keywords: oxidative stress, antioxidant, periodontitis, serum immunoglobulin G; antibody titer
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Nagasaki: Sample collection
- Tokushima: Oxidative stress, cytokine
- Kanagawa: oxidative stress

SUMMARY:
we analyzed the relationship between oxidative stress, immunoglobulin G antibody titers, cytokines, and periodontitis through community-based study held in the Goto city, Japan.

ELIGIBILITY:
Inclusion Criteria:

more than 15 teeth

Exclusion Criteria:

less than 15 teeth

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-03 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
oxidative stress and periodontitis | participants will be followed by an expected average of 1 year.
  reactive oxygen metabolites were measured. immunoglobulin G antibodies were measured by enzyme-linked immunosorbent assay.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nagasaki, Nagasaki, Goto, Japan

REFERENCES:
- [Background] Hayashida H, Kawasaki K, Yoshimura A, Kitamura M, Furugen R, Nakazato M, Takamura N, Hara Y, Maeda T, Saito T. Relationship between periodontal status and HbA1c in nondiabetics. J Public Health Dent. 2009 Summer;69(3):204-6. doi: 10.1111/j.1752-7325.2009.00122.x. PMID 19486462
- [Derived] Tamaki N, Yoshino F, Fukui M, Hayashida H, Yoshida A, Kitamura M, Iwasaki T, Furugen R, Kawasaki K, Nakazato M, Maeda T, Kokeguchi S, Yamamoto T, Lee MC, Ito HO, Saito T. Relationship among salivary antioxidant activity, cytokines, and periodontitis: the Nagasaki Island study. J Clin Periodontol. 2015 Aug;42(8):711-718. doi: 10.1111/jcpe.12438. Epub 2015 Aug 29. PMID 26227009
- See also: Japanese — http://www.mh.nagasaki-u.ac.jp/soshin/index.html